CLINICAL TRIAL: NCT04439136
Title: MATCH Treatment Subprotocol B: Phase II Study of Afatinib in Patients With Tumors With HER2 Activating Mutations
Brief Title: Testing Afatinib as a Potential Targeted Treatment in Cancers With HER2 Genetic Changes (MATCH-Subprotocol B)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2020-03140; NCI-2020-03140 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EAY131-B (Other: ECOG-ACRIN Cancer Research Group); EAY131-B (Other: CTEP); U10CA180820 (NIH); U24CA196172 (NIH)
Record Dates: First submitted 2020-06-18; First posted 2020-06-19 (Actual); Results first posted 2022-11-29 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Advanced Lymphoma; Advanced Malignant Solid Neoplasm; Hematopoietic and Lymphoid Cell Neoplasm; Refractory Lymphoma; Refractory Malignant Solid Neoplasm; Refractory Multiple Myeloma
MeSH Terms: conditions — Hematologic Neoplasms; Lymphoma; Multiple Myeloma | interventions — Afatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (afatinib dimaleate) (Experimental): Patients receive afatinib dimaleate PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Afatinib Dimaleate

INTERVENTIONS:
Drug: Afatinib Dimaleate — Given PO
  Other Names: (2E)-N-(4-((3-Chloro-4-fluorophenyl)amino)-7-(((3S)-tetrahydrofuran-3-yl)oxy)quinazolin- 6-yl)-4-(dimethylamino)but-2-enamide bis(hydrogen (2Z)-but-2-enedioate); BIBW 2992MA2; BIBW2992 MA2; Gilotrif

SUMMARY:
This phase II MATCH treatment trial identifies the effects of afatinib in patients whose cancer has genetic changes called HER2 mutations. Afatinib may stop the growth of cancer cells by blocking the HER2 receptor, a protein that may be needed for cell growth. Researchers hope to learn if afatinib will shrink this type of cancer or stop its growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the proportion of patients with objective response (OR) to targeted study agent(s) in patients with advanced refractory cancers/lymphomas/multiple myeloma.

SECONDARY OBJECTIVES:

I. To evaluate the proportion of patients alive and progression free at 6 months of treatment with targeted study agent in patients with advanced refractory cancers/lymphomas/multiple myeloma.

II. To evaluate time until death or disease progression. III. To identify potential predictive biomarkers beyond the genomic alteration by which treatment is assigned or resistance mechanisms using additional genomic, ribonucleic acid (RNA), protein and imaging-based assessment platforms.

IV. To assess whether radiomic phenotypes obtained from pre-treatment imaging and changes from pre- through post-therapy imaging can predict objective response and progression free survival and to evaluate the association between pre-treatment radiomic phenotypes and targeted gene mutation patterns of tumor biopsy specimens.

OUTLINE:

Patients receive afatinib dimaleate (afatinib) orally (PO) once daily (QD) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months if less than 2 years from study entry, and then every 6 months for year 3 from study entry.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have met applicable eligibility criteria in the Master MATCH Protocol prior to registration to treatment subprotocol
* Patient's tumor must have activating HER2 mutation, as determined via the MATCH Master Protocol

  * Additionally, any in-frame insertions in exon 20 will be considered an activating mutation
* Patients must have an electrocardiogram (ECG) within 8 weeks prior to treatment assignment and must have no clinically important abnormalities in rhythm, conduction or morphology of resting ECG (e.g. complete left bundle branch block, third degree heart block)
* Patients with known left ventricular dysfunction must have echocardiogram (ECHO) or a nuclear study (multiple-gated acquisition [MUGA] or First Pass) within 4 weeks prior to registration to treatment and must not have left ventricular ejection fraction (LVEF) < institutional lower limit of normal (LLN). If the LLN is not defined at a site, the LVEF must be > 50% for the patient to be eligible

  * NOTE: Pre-treatment LVEF determination in patients without known left ventricular dysfunction is NOT otherwise required.
* Patients must have =< grade 1 diarrhea at baseline
* Patients must have =< grade 1 renal function as defined below:

  * Creatinine =< 1.5 x normal institutional limits OR
  * Measured creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal or as calculated by the Cockcroft-Gault equation

    * This should be strictly followed and will override the MATCH Master Protocol requirements

Exclusion Criteria:

* Patients must not have known hypersensitivity to afatinib or compounds of similar chemical or biologic composition
* Patients with a history of interstitial lung disease will be excluded
* Patients must not have had prior treatment with any of the following tyrosine kinase inhibitors (TKIs), which have known activity against HER2 kinase:

  * Neratinib
  * AC-480 (BMS-599626)
  * AST 1306
  * Canertinib (CI 1033)
  * CUDC-101
  * Lapatinib
  * TAK285
  * Afatinib
  * AEE 788
  * AZD8931
  * CP-724714
  * Dacomitinib
  * Pelitinib
* Patients with non-small cell lung cancer will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-08-12 (Actual); Primary Completion 2021-01-22 (Actual); Study Completion 2026-03-17 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe L Bedard, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (1):
- ECOG-ACRIN Cancer Research Group, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subprotocol B was activated on August 12, 2015. Fifty-nine patients were assigned to Subprotocol B after screening, all from screening cohort. Of the 59 patients, 40 patients were enrolled in arm B between August 2015 and June 2017.
Pre-assignment Details: To be assigned to a specific MATCH subprotocol, patients needed to submit a tumor biopsy for molecular characterization and those with molecular variants addressed by treatments included in the trial entered corresponding MATCH subprotocol. For the subprotocol B, patients had to have a qualifying ERBB2 actionable mutation.
Groups:
- Treatment (Afatinib Dimaleate): Patients receive afatinib dimaleate 40mg PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Afatinib Dimaleate: Given PO
Period: Overall Study
Arm/Group | Treatment (Afatinib Dimaleate)
Started | 40
Eligible | 39
Eligible and Started Protocol Therapy (One patient ineligible, 2 patients never started treatment. This is the primary analysis population.) | 37
Reported Adverse Events Data (Excluding two who did not receive afatinib treatment and one who was not assessed for toxicity) | 37
Completed (Treatment continued until disease progression or intolerability.) | 0
Not Completed | 40
Not completed — Ineligible | 1
Not completed — Never Started Treatment | 2
Not completed — Adverse Event | 4
Not completed — Death | 3
Not completed — Disease Progression | 27
Not completed — Alternative Therapy | 1
Not completed — Increased Tumor Burden | 1
Not completed — Symptomatic Detrioration | 1

BASELINE CHARACTERISTICS:
Population: Eligible and treated patients
Arm/Group | Treatment (Afatinib Dimaleate)
Number analyzed (Participants) | 37
Age, Continuous [Median (Full Range); unit: years] | 62 [29 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 30
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: Overall response rate was defined as the proportion of patients with best overall response of complete response (CR) or partial response (PR) among all eligible and treated patients. Best overall response was evaluated using the Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. Please refer to the protocol for the detailed definitions of response criteria. The 90% two-sided binomial exact confidence interval was calculated for ORR.
Time Frame: Tumor assessments occurred at baseline, then every 2 cycles for the first 26 cycles and every 3 cycles thereafter until disease progression, up to 3 years post registration
Population: Patients who were eligible and received protocol treatment
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Afatinib Dimaleate)
Number analyzed (Participants) | 37
percentage of participants | 2.7 [0.14 to 12.2]

2. Secondary Outcome: 6-month Progression-free Survival (PFS) Rate
Description: Progression free survival is defined as time from treatment start date to date of progression or death from any cause, whichever occurs first. Disease progression was evaluated using the Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. Please refer to the protocol for detailed definitions of disease progression. 6 month PFS rate was estimated using the Kaplan-Meier method, which can provide a point estimate for any specific time point.
Time Frame: Assessed at baseline, then every 2 cycles for the first 26 cycles, and every 3 cycles thereafter until disease progression, up to 3 years post registration, from which 6-month PFS rate is determined
Population: Patients who were eligible and received protocol treatment
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Afatinib Dimaleate)
Number analyzed (Participants) | 37
percentage of participants | 12.0 [5.6 to 25.8]

3. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as time from treatment start date to date of disease progression or death from any causes, whichever occurred first. Median PFS was estimated using the Kaplan-Meier method. Disease progression was evaluated using the Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. Please refer to the protocol for detailed definitions of disease progression.
Time Frame: Assessed at baseline, then every 2 cycles for the first 26 cycles and every 3 cycles thereafter until disease progression, up to 3 years post registration
Population: Patients who were eligible and received protocol treatment
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Treatment (Afatinib Dimaleate)
Number analyzed (Participants) | 37
months | 1.7 [1.6 to 4.2]

ADVERSE EVENTS:
Time Frame: Assessed every 28 days while on treatment and for 30 days after the end of treatment, up to 3 years post registration.
Description: All patients enrolled were included in the all-cause mortality analysis. Thirty-seven patients were included in the toxicity analysis (excluding two who did not receive afatinib treatment and one who was not assessed for toxicity).
Arm/Group | Treatment (Afatinib Dimaleate)
All-Cause Mortality (participants affected / at risk) | 37/40
Serious Adverse Events (participants affected / at risk) | 18/37
Other Adverse Events (participants affected / at risk) | 31/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Afatinib Dimaleate) (N=37)
Anemia (Blood and lymphatic system disorders) | 2
Fatigue (General disorders) | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Anal hemorrhage (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 7
Mucositis oral (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 1
Sepsis (Infections and infestations) | 2
Alkaline phosphatase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 2
Creatinine increased (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 1
White blood cell decreased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Afatinib Dimaleate) (N=37)
Anemia (Blood and lymphatic system disorders) | 8
Chills (General disorders) | 2
Fatigue (General disorders) | 13
Fever (General disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 3
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 4
Rash acneiform (Skin and subcutaneous tissue disorders) | 11
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 3
Constipation (Gastrointestinal disorders) | 5
Diarrhea (Gastrointestinal disorders) | 24
Dry mouth (Gastrointestinal disorders) | 5
Mucositis oral (Gastrointestinal disorders) | 13
Nausea (Gastrointestinal disorders) | 10
Vomiting (Gastrointestinal disorders) | 10
Paronychia (Infections and infestations) | 2
Alanine aminotransferase increased (Investigations) | 4
Alkaline phosphatase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 4
Creatinine increased (Investigations) | 2
Lymphocyte count decreased (Investigations) | 3
Platelet count decreased (Investigations) | 2
Weight loss (Investigations) | 4
White blood cell decreased (Investigations) | 2
Investigations - Other, specify (Investigations) | 2
Anorexia (Metabolism and nutrition disorders) | 7
Dehydration (Metabolism and nutrition disorders) | 9
Hypoalbuminemia (Metabolism and nutrition disorders) | 3
Hypokalemia (Metabolism and nutrition disorders) | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 4
Hyponatremia (Metabolism and nutrition disorders) | 3
Musculoskeletal and connective tissue disorder - Other, spe (Musculoskeletal and connective tissue disorders) | 2
Dysgeusia (Nervous system disorders) | 3
Blurred vision (Eye disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol (2019-07-10): https://cdn.clinicaltrials.gov/large-docs/36/NCT04439136/Prot_001.pdf